CLINICAL TRIAL: NCT06537596
Title: An Open-label, Phase 1 Study to Assess Safety, Tolerability, Dosimetry, Pharmacokinetics and Imaging Properties of 89Zr-olaratumab (89Zr-TLX300-CDx) in Participants With Soft Tissue Sarcoma.
Brief Title: 89Zr-olaratumab Dosimetry in Participants With Soft Tissue Sarcoma
Acronym: ZOLAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 89Zr-TLX300-101
Record Dates: First submitted 2024-04-29; First posted 2024-08-05 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Proof-of-concept tumour targeting of 89Zr-TLX300-CDx (Part A), assessment of 89Zr-TLX300-CDx biodistribution and tumour uptake (Part B) and radiation dosimetry (Part C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): One Injection of 89Zr-TLX300-CDx
  Interventions: Drug: 89Zr-DFOsq-olaratumab (89Zr-TLX300-CDx)
- Part B (Experimental): One Injection of 89Zr-TLX300-CDx
  Interventions: Drug: 89Zr-DFOsq-olaratumab (89Zr-TLX300-CDx)
- Part C (Experimental): One Injection of 89Zr-TLX300-CDx
  Interventions: Drug: 89Zr-DFOsq-olaratumab (89Zr-TLX300-CDx)

INTERVENTIONS:
Drug: 89Zr-DFOsq-olaratumab (89Zr-TLX300-CDx) — Single administration of 89Zr-TLX300-CDx

SUMMARY:
Soft Tissue Sarcoma (STS) is a type of cancer that develops in soft tissues such as muscles, tendons, fat, blood vessels, and nerves. STSs generally express a protein called Platelet-Derived Growth Factor Receptor (PDGFR)α, which makes them a target for the development of STS therapies, such as olaratumab.

Olaratumab has been identified as a promising candidate to which radioactive substances can be attached for imaging or therapeutic purposes. Thus, this first in human imaging trial aims to study olaratumab combined with a radioactive metal called zirconium-89 (89Zr-TLX300-CDx) as a potential new product that may be used for STS imaging and identification of patients that may benefit from future treatments targeting PDGFRα.

DETAILED DESCRIPTION:
Platelet-derived growth factor receptor α (PDGFRα) is expressed on soft tissue sarcoma (STS) where it could act as a potential therapeutic target. Olaratumab is a PDGFRα-targeted antibody that has the potential to act as the targeting moiety for both imaging and therapeutic radioisotopes. Olaratumab's demonstrated safety profile and its ability to target PDGFRα on STS cell surfaces and be rapidly internalised, make it a promising candidate for use as a radionuclide targeting agent in STS. 89Zr-TLX300-CDx is being developed for PDGFRα molecular imaging with positron emission tomography (PET) in STS. The aim of this study is to provide proof-of-concept tumour targeting of 89Zr-TLX300-CDx and assess the safety and radiation dosimetry of radiolabelled olaratumab. This study will inform future development of olaratumab as a therapeutic radiopharmaceutical agent in STS.

SCHEDULE OF ASSESSMENTS

Part A and B:

IMAGING:

1 single injection of 89Zr-TLX300-CDx on Day 1 and whole-body imaging at 6 days ± 1 day post-injection

Blood Collection for PHARMACOKINETICS:

Pre-injection, 4h ± 0.5h and 6 days ± 1 day post-injection.

OPTIONAL:

Imaging at 4h ± 0.5h post-injection.

Part C:

IMAGING:

1 single injection of 89Zr-TLX300-CDx on Day 1, whole-body imaging at 24h ± 4h post-injection, whole-body imaging at 4 days ± 1 post-injection and whole-body imaging at 7 days ± 1 day post-injection

Blood collection for PHARMACOKINECTCS:

Pre-injection, 4h ± 0.5h, 24h ± 4h, 4 days ± 1 day and 7 days ± 1 day post-injection.

OPTIONAL:

Dynamic imaging 15 min ± 2 min post-injection at selected sites (extended field-of-view scanner is available), imaging at 4h ± 0.5h post-injection and imaging at 7h ± 1hpost-injection

ELIGIBILITY:
INCLUSION CRITERIA:

1. ≥18 years of age at the time of signing the informed consent.
2. Histologically confirmed diagnosis of soft tissue sarcoma (STS)
3. At least one mass of > 2 cm in largest diameter seen on standard of care imaging (CT, MRI and/or FDG-PET).
4. For Part A: Participants must have tumour PDGFRα expression confirmed by IHC. Participants must have consented to provide archived FFPE tumour tissue or be subject to a biopsy of the target tumour (if archived tissue is unavailable).

   For Parts B and C: all participants will be included regardless of their PDGFRα expression status on archival tissue/biopsy (unless otherwise specified). Participants must have consented to provide available archived FFPE tumour tissue.
5. Adequate haematologic function as defined by an absolute neutrophil count (ANC) ≥ 1500/ μL, haemoglobin ≥ 9.0 g/dL, and a platelet count of 100,000/μL obtained.
6. Adequate hepatic function as defined by a total bilirubin ≤ 1.5 mg/dL, and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (ULN).
7. Adequate renal function as defined by serum creatinine ≤ 1.5 × the institutional ULN. If creatinine is above the ULN, the participant's creatinine clearance is ≥ 45 mL/min.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
9. Life expectancy of at least 6 months.
10. Female participants of childbearing potential must have negative pregnancy tests at screening, as well as confirmation of negative pregnancy test result within 24 hours prior to receiving 89Zr-TLX300-CDx. Female participants of childbearing potential or male participants with female partners of childbearing potential must:

    1. be willing to practice full and true sexual abstinence; or
    2. be surgically/permanently sterile or with a history of hysterectomy for women; or
    3. be willing to practice highly effective contraception by using: a non-oral, injected or implanted non-oestrogen progesterone based hormonal method, male condom, vaginal diaphragm, cervical cap, intrauterine device, for 3 months after the administration of 89Zr-TLX300-CDx.
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

EXCLUSION CRITERIA:

1. Known or suspected hypersensitivity to olaratumab, DFOsq, 89Zr or any of the excipients.
2. IgE antibodies against galactose-α-1,3-galactose (α-Gal) above the upper limit of normal, > 0.7 kU/L.
3. Exposure to any experimental diagnostic or therapeutic drug within 30 days from the date of planned administration of 89Zr-TLX300-CDx.
4. Surgery ≤ 2 weeks prior to the administration of 89Zr-TLX300-CDx or significant ongoing complications of surgery. Biopsy ≤ 2 weeks prior to the administration of 89Zr-TLX300-CDx is allowed.
5. Exposure to any radiopharmaceutical within 10 half-lives prior to the administration of 89Zr-TLX300-CDx.
6. Ongoing toxicity Grade 2 or higher from previous standard or investigational therapies (Common Terminology Criteria for Adverse Events [CTCAE] version 5).
7. Planned to commence systemic antineoplastic therapies, immunotherapy, targeted therapy, radiotherapy and/or surgery for the period between administration of 89Zr-TLX300-CDx and last imaging timepoint.
8. Serious non-malignant disease (e.g., psychiatric, infectious, autoimmune or metabolic) or any disease that may interfere with the objectives of the study or with the safety or compliance of the participant, as judged by the Investigator.
9. Pregnant or lactating women.
10. Participants unable to declare meaningful informed consent on their own (e.g., with legal guardian for mental disorders) or unable to tolerate the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate clinical safety and tolerability of 89Zr-TLX300-CDx | 30 days
  Number of Adverse events (AEs)
Biodistribution of 89Zr-TLX300-CDx | 6 days
  Measurement of absorbed radiation doses to organs.
Radiation dosimetry of 89Zr-TLX300-CDx | 6 days
  Measurement of absorbed radiation doses to tumour(s) and whole body.
Pharmacokinetics (PK) | 6 days
  Measure the antibody concentration at each timepoint to determine a PK curve.

SECONDARY OUTCOMES:
Determine a suitable antibody mass for administration | 6 days
  SUV values of tumour lesions and tumour to background organ (e.g. blood/liver/muscle) ratios.

OTHER OUTCOMES:
Evaluate the correlation between tumour uptake of 89Zr-TLX300-CDx and PDGFRα expression | 30 days
  Immunohistochemistry expression of PDGFRα in tumour tissue AND SUV tumour values and tumour to background ratios.
Compare the tumour uptake and detection of lesions between 89Zr-TLX300-CDx and standard of care imaging | 30 days
  89Zr-TLX300-CDx uptake within tumours and organs and Localisation of tumour deposits on conventional imaging (CT, MRI and/or FDGPET)

CONTACTS AND LOCATIONS:
Locations (1):
- Precision Molecular Imaging & Theranostics Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No